CLINICAL TRIAL: NCT05848791
Title: Respiratory Impacts of Tailpipe and Non-tailpipe Particulates on Adults With Asthma: A Feasibility Study
Brief Title: Assessing the Impact of Non-tailpipe Emissions From Traffic on the Asthmatic Airway
Acronym: IONA
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Asthma UK (Other); Health Effects Institute (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, James Scales, Research Fellow (AUKCAR), Queen Mary University of London
Other Study IDs: 320784; 156019 (Other: EDGE Number); 55343 (Other: CPMS Number); AUK-AC-2018 (Other Grant/Funding Number: Asthma and Lung UK Centre for Applied Research); CR-83590201 (Other: Health Effects Instutute)
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Plasma. Nasal Mucus. Urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise exposure — Participants are exposed to three different air quality environments in central London, chosen to maximise differences in nontailpipe air pollution. Participants will cycle at 60% of estimated maximum vo2 on static bikes for six 15 minute bouts with 15 minutes rest between bouts.

SUMMARY:
The goal of this observational study is to explore the health impacts of exposure to nontailpipe vehicle air pollution. The main question it aims to answer is: Does short term exposure to increased non-tailpipe course mode PM induce negative respiratory responses in adults living with asthma?

We will recruit 48 non-smoking adults with mild-moderate asthma. Participants will be recruited from central and east London

Participants will be exposed to three contrasting air quality environments, in field laboratories at the following locations:

1. High-speed continuous traffic location, to enhance tire wear emissions
2. An urban background location away from nearby traffic sources
3. A busy road junction characterized by stop-go traffic to enhance emissions from brake wear

Sites 1 and 2 are permanent air quality measurement supersites. Site 1 is located close to a major trunk road in Central London (Marylebone Road). Site 2 is a suburban park in South London (Honor Oak Park). An additional measurement location will be established at Imperial College London's (ICL) White City campus (Site 3) for the duration of the study using ICL's mobile measurement facility, equipped with the same highly time-resolved chemical composition measurement capability as the supersites.

To maximise exposure to different air quality environments participants will intermittently cycle on static exercise bikes at a standardised intensity of 60% estimated VO2max for a duration for 2.5 hours at the field laboratories.

Comparators variables:

Air quality will be monitored at all three sites for the duration of the testing visits (approximately 5 hours). Air quality parameters that will be recorded are PM2.5, PM10, NO2, NO, NOX, O3, Organic Mass, NO3, SO4, NH4, elements and black carbon.

Outcome variables:

The primary outcome of the study is lung function as measured by Forced Expiratory Volume in one second (FEV1). With secondary health endpoints including: Spirometry (FVC, FVC/FEV1 ratio, z Scores), fractional expired nitric oxide (FeNO), oscillometry, asthma symptoms, MRC breathlessness score, asthma control test and Asthma Quality of Life Questionnaire (AQLQ). Blood, nasal mucus and urine samples will be collected. Measure will be collected before after and 24 hours after exposure.

DETAILED DESCRIPTION:
Participants will be invited to take part by either Dr James Scales or by a primary care practitioner in their General Practice clinics. Participants will provide informed consent after they have read the study information sheets and have time consider their involvement (minimum 24 hours) and ask any questions.

Upon providing informed consent the participants will visit QMUL laboratories for a screening assessment. During this one hour visit they will complete a submaximal exercise test on a static bike (to provide estimates of maximal exercise capacity to standardise exercise exposure protocol) and perform pre and post bronchodilator spirometry and exhaled nitric oxide testing and oscillometry. At this point participants will be sent an online link to the symptom surveys. Surveys will be explained to the participants and they will be asked to complete the surveys they days before the testing visits. Participants will be provided with personal air quality monitor, heart rate monitor and physical activity monitor to wear three days before the exposure visit.

Participants will be invited to visit one of three field based study sites in a random order. Study sites will be located in walled gazebos next to air quality monitoring sites (managed by our collaborators at ICL) positioned near roads to provide the required air quality exposure. The protocol for the three visits will be identical and each visit will be separated by at least two weeks (washout). Participants will initially provide a urine sample at home and will bring the sample with them to the testing site. To control for participant exposures before testing, a taxi will be provided for the participant. Participants will travel with car windows closed, and air recirculation turned on. Participants will arrive that the study site at 10:00am, and will be joined by up to three other participants. In the first hour the participants will perform the respiratory health assessments and will provide a blood and a nasal mucus sample. After performing all the pre exercise tests participants will wear a heart rate monitor and will commence the exercise protocol (six exercise bouts of 15 minutes separated by fifteen-minute rest periods on a static exercise bike). Half-way through the protocol participants will perform spirometry, impulse oscillometry and FeNO testing. Upon completing the two-hour exercise protocol participants will complete the same battery of health assessments and will provide nasal mucus samples. Participants will leave the assessment area at about 14:00pm. Air pollution measurements will be taken for the duration of the time that the participant visits the exercise location.

24 hours after the exercise protocol participants will visit the QMUL laboratories to perform the health assessment tests again and to provide a mucus sample via nasal lavage, blood sample via venepuncture and provide a urine sample. After repeating this process three times (one visit to each field site) they will receive an expenses payment of £200 and leave the study. Participants will be paid £60 per exposure visit and £20 pre-screening visit. Participants will be paid for each visit they attend and will be paid when they complete participation or withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma starting on or before age 16 years
* Prescribed regular inhaled corticosteroid medication
* Able to use a static exercise bicycle for the study duration

Exclusion Criteria:

* Tobacco smoking, or living with smoker
* Body mass index (BMI) > 30
* Asthma hospitalisation within 12 months
* Three or more asthma episodes requiring oral corticosteroid medication within 12 months
* Other major lung disease
* Chest surgery within 6 months
* Unable to give informed consent
* Occupational exposure to particulate matter (PM) or high levels of air pollution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from universities and general practices in London.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory volume in one Second (FEV1) | 0 hours and 2.5hours.
  FEV1 as measured by spirometry

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | 0 hours, 2.5hours and 26 hours
  FVC as measured by spirometry
Change in Fractional expired Nitric Oxide | 0 hours, 2.5hours and 26 hours
  (FeNO)
Change in Daily asthma symptoms | 0 hours, 2.5hours and 26 hours
  Via validated questionaire
Change in Immune response | 0 hours, 2.5hours and 26 hours
  damage-associated molecular patterns (DAMPs) and alarmins, such as high mobility group box 1 (HMGB1) S100 proteins, myeloperoxidase-DNA complexes (MPO-DNA), IL-33, Th2 and Th17 cytokines and metal deposition in the nasal airways
Change in Airway resistance | 0 hours, 2.5hours and 26 hours
  Airway resistance as measured by impulse oscillometry

CONTACTS AND LOCATIONS:
Overall Officials: James Scales, PhD, Principal Investigator — Queen Mary University London
Locations (1):
- Queen Mary University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT05848791/Prot_000.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT05848791/ICF_001.pdf